CLINICAL TRIAL: NCT05514782
Title: Double-Blinded, Placebo-Controlled, Randomized Study to Evaluate the Efficacy and Tolerability of a Daily Serum
Brief Title: A Clinical Study to Evaluate the Long-Term Efficacy and Tolerability of a Daily Anti-Aging Daily Serum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Collaborators: KGL, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 8602
Record Dates: First submitted 2022-08-17; First posted 2022-08-24 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Photoaging; Wrinkle
Keywords: anti-aging; daily serum
MeSH Terms: interventions — cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, single-center
Who Masked: Participant, Investigator
Masking Description: Randomization occurred by assignment to either Cell 1 or Cell 2 using a randomization list, prepared by KGL Skin prior to the start of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-Aging Daily Serum (Active Comparator): Daily serum composed of a patent-pending botanical extract, bioavailable peptide, antioxidants, postbiotic(s), short term and long-term moisturizers. New product in development.
  Interventions: Other: Cleansing Lotion; Other: Facial Moisturizer; Other: Sunscreen SPF 40+
- Placebo-Control (Placebo Comparator): Vehicle control of the anti-aging daily serum.
  Interventions: Other: Cleansing Lotion; Other: Facial Moisturizer; Other: Sunscreen SPF 40+

INTERVENTIONS:
Other: Cleansing Lotion — Facial cleansing lotion to be used by study participants (morning and evening, 2x daily).
  Other Names: Revision Skincare® Cleansing Lotion
Other: Facial Moisturizer — Anti-aging facial moisturizer to be used by study participants after anti-aging daily serum before sunscreen.
  Other Names: Goodier Cosmetics Facial Moisturizer
Other: Sunscreen SPF 40+ — Sunscreen to be applied after application of the facial moisturizer in the morning. Participants were asked to reapply every 2 hours.
  Per FDA this intervention is an Over the counter
  Other Names: Aveeno Positively Mineral Sensitive Skin SPF 40+)

SUMMARY:
This double-blind, randomized, placebo-controlled, single-center clinical trial was conducted to assess the efficacy and tolerance of an anti-aging daily serum to improve moderate overall photodamage and skin fatigue after 12-weeks of twice-daily used when compared to a placebo-serum (vehicle control). A total of 62 subjects, 34-60 years of age completed study participation.

DETAILED DESCRIPTION:
This double-blind, randomized, placebo-controlled, single-center clinical trial was conducted to assess the efficacy and tolerance of an anti-aging daily serum (Cell 1) to improve moderate overall photodamage and skin fatigue of aging skin after 12-weeks days of twice-daily use when compared to the efficacy of a combination of a placebo-control (Cell 2). Skin fatigue was characterized by dehydrated skin with a lack of firmness (visual) and a dull appearance on the global face.

Efficacy and tolerability were assessed through clinical grading at baseline, week 4, week 8, and week 12. Efficacy evaluation on fine lines and wrinkles in the crow's feet area; overall eye appearance on the periocular area; and smoothness (tactile), firmness (visual), radiance, and overall photodamage on the global face were performed at baseline and post-baseline by a clinical grader, a board-certified dermatologist. Furthermore, blinded photo-grading at baseline and week 12 were performed by two board certified dermatologists.

Self-assessment questionnaires, Antera 3D image, Ultrasound Imaging, and VISIA photography were completed at baseline and post-baseline timepoints. Furthermore, 10 randomized subjects, a subset of the study (five in Cell 1 and five in Cell 2) had 2 mm punch skin biopsies collected from the lateral, pre-auricular at baseline and week 12.

A total of 62 subjects completed study participation (31 in Cell 1 and 31 in Cell 2).

ELIGIBILITY:
Inclusion Criteria:

* Female 30 to 60 years of age
* Fitzpatrick skin type I -IV
* Moderate overall photodamage of the skin
* Moderate lack of firmness (visual) of the skin
* Moderate dull appearance of the skin
* Subjects must be willing to withhold all facial treatments during the course of the study and have not undergone a treatment within the last 6 months
* Subject must be willing to provide verbal understanding and written informed consent

Exclusion Criteria:

* Diagnosed with known allergies to facial skincare products
* Nursing, pregnant, or planning to become during the duration of the study
* History of skin cancer within the past 5 years
* Having used oral isotretinoin within the last 12 months
* Having used prescription-strength skin-lightening products within the last 3 months
* Having used any anti-wrinkle, skin-lightening, or other product or topical or systemic medication known to affect skin aging or dyschromia within the last 4 weeks
* Having a health condition and/or pre-existing or dermatologic disorder that, in the Investigator's opinion, may interfere with the outcome of the study
* Having observable sunburn, suntan, scars, excessive facial hair, or other dermal conditions on the face that, in the Investigator's opinion, may influence test results
* Having a history of immunosuppression/immune deficiency disorders, or currently using oral or systemic immunosuppressive medications and biologics, and/or undergoing radiation or chemotherapy
* Using or having regularly used systemic or topical corticosteroids within the past 4 weeks
* Having started a long-term medication within the last 2 months

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Change In Clinical Efficacy Parameter Radiance Versus Baseline | 12 weeks
  The primary efficacy endpoint will be the Investigator Clinical Grading using Modified Griffith's 10-point Scale at post-baseline timepoints.
  A decrease in scores at post-baseline timepoints (week 4,8, and12) in comparison to baseline indicates an improvement for the indicated parameter.
  The efficacy parameters will be assessed globally on each subject's face using a modified Griffiths' 10-point scale according to the following numerical definitions (half-point scores may be used as necessary to more accurately describe the skin condition):
  0 = none (best possible condition); 1 to 3 = mild; 4 to 6 = moderate;7 to 9
  = severe (worst possible condition). The lower the score equates to the best possible outcome.
Change in Active Cell versus Placebo Control in Clinical Efficacy at week 12 | 12 weeks
  The primary efficacy endpoint will be the Investigator Clinical Grading using Modified Griffith's 10-point Scale at post-baseline timepoints versus the placebo control.
  A confidence interval of 90% (p <0.10) for both live clinical grading and photo-grading will be performed between the Cell 1 (active comparator) versus Cell 2 (placebo control comparator).
  The efficacy parameters will be assessed globally on each subject's face using a modified Griffiths' 10-point scale according to the following numerical definitions (half-point scores may be used as necessary to more accurately describe the skin condition):
  0 = none (best possible condition); 1 to 3 = mild; 4 to 6 = moderate;7 to 9
  = severe (worst possible condition). The lower the score equates to the best possible outcome.

SECONDARY OUTCOMES:
Lack of Significant Increase in Objective Investigator Tolerability Parameters at week 4, 8, 12 compared to Baseline | 12 weeks
  The second outcome measure is objective tolerability endpoint. Investigator Tolerability Assessment includes Erythema, Edema and Dryness.
  A decrease in scores or lack of significant increase at week 4, 8, and 12 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example for Erythema: Erythema 0 = None No erythema of the treatment area
  1. = Mild Slight, but definite redness of the treatment area
  2. = Moderate Definite redness of the treatment area
  3. = Severe Marked redness of the treatment area
Lack of Significant Increase in Subjective Tolerability Parameters at week 4, 8, 12 compared to Baseline | 12 weeks
  The secondary tolerability endpoint will be the Subjective Tolerability Assessment of Burning, Itching and Stinging.
  A decrease in scores or lack of significant increase at week 4, 8, and 12 in comparison to Baseline indicates tolerability/safety of the test material. Four point scale with a lower score indicating a better outcome.
  Example Burning. 0 = None No burning of the treatment area
  1. = Mild Slight burning sensation of the treatment area; not really bothersome
  2. = Moderate Definite warm, burning of the treatment area that is somewhat bothersome.
  3. = Severe Hot burning sensation of the treatment area that causes definite discomfort and may interrupt daily activities and/or sleep

OTHER OUTCOMES:
Change In Facial parameters in a self-assessment questionnaire versus Baseline and % Agreement | 12 weeks
  Self-Assessment Questionnaire and the Subject Treatment Satisfaction. A decrease or increase in response values at week 4, 8, and 12, and indicates an improvement compared to baseline response values.
  Subjects are asked to rate based on a scoring system of the following:
  from 5 (completely agree) to 1 (completely disagree). The best outcome is to Completely Agree with the statement/ question being asked.
Bioinstrumentation -Quantitative and Qualitative Data | 12 weeks
  Bioinstrumentation measurements includes Antera 3D imaging (Miravex Limited, Dublin, Ireland).
  Measurements are taken of either the right or left cheek area at baseline, week 8 and week 12. Comparisons are made to baseline.
  A decrease in skin redness and skin melanin pigmentation indicates an improvement.
Bioinstrumentation - Quantitative and Qualitative Data | 12 weeks
  Bioinstrumentation measurements includes Ultrasound Imaging (DermaScan C; Cortex Technology, Hadsund, Denmark). Measurements are taken of either the right or left cheek area at baseline, week 8 and week 12. Comparisons are made to baseline.
  An increase in skin density over time indicates improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- KGL Skin Study Center, West Chester, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No